CLINICAL TRIAL: NCT04383535
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial of Convalescent Plasma for the Treatment of COVID-19 Pneumonia With Severity Criteria
Brief Title: Convalescent Plasma and Placebo for the Treatment of COVID-19 Severe Pneumonia
Acronym: PLASM-AR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5565
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: SARS Virus; SARS-CoV-2; COVID-19
Keywords: SARS Virus; SARS-CoV-2; COVID-19; Blood Plasma
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: Multicenter randomized (2:1, 222 plasma 111 placebo), double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacist will be unblinded. The study intervention will be covered with an opaque development in order to ensure blinding of the intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent SARS COVID-19 plasma (Experimental): Convalescent SARS COVID-19 plasma from a pool of 10 donor plasma, in addition to standard care.
  Interventions: Other: Convalescent SARS COVID-19 plasma
- Placebo (Placebo Comparator): Single infusion of saline solution, in addition to standard care.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Convalescent SARS COVID-19 plasma — Convalescent SARS COVID-19 plasma from a pool of 10 donor plasma. The calculation of the volume to be transfused will be from 10 to 15 ml / kg adjusting the volume to the body weight of each patient, at a suggested infusion rate of 5 to 10 ml / kg / h with an intravenous infusion pump. The infusion rate will be adjusted according to the clinical stability of the patient according to the treating physician.
  Arms: Convalescent SARS COVID-19 plasma
Other: Placebo — Single infusion of saline solution, in addition to standard care. The calculation of the volume to be transfused will be from 10 to 15 ml / kg adjusting the volume to the body weight of each patient, at a suggested infusion rate of 5 to 10 ml / kg / h with an intravenous infusion pump. The infusion rate will be adjusted according to the clinical stability of the patient according to the treating physician.
  Arms: Placebo

SUMMARY:
A multicenter randomized, double-blind, placebo-controlled clinical trial of Convalescent SARS COVID-19 plasma versus Placebo to evaluate the effect between arms on an ordinal score of six mutually exclusive categories of clinical status at day 30 after study initiation.

DETAILED DESCRIPTION:
Introduction

The use of convalescent plasma in the treatment of infectious diseases has been empirically performed for more than a century. It is based upon the assumption that providing exogenous neutralizing antibodies may provide protection while affected patients mount their own immune response. This therapeutic approach appears of particular interest in the context of the current pandemic, in which there is no specific vaccine available nor adequately proven effective pharmacological treatments.

Study purpose, hypothesis and general design

Purpose of the study: evaluate the effectiveness and safety of convalescent plasma in the treatment of SARS-CoV-2 pneumonia (Covid-19) Hypothesis: Convalescent plasma significantly improves the clinical outcome in patients with Covid-19 pneumonia and severity criteria.

Multicenter randomized, double-blind, placebo.controlled clinical trial. Placebo will be a saline solution.

3. Methodological sustain for including a control arm with placebo Quality evidence about the effectiveness of convalescent plasma in the treatment of Covid-19 pneumonia is not yet available. Although case series and anecdotal reports appear encouraging, the implementation of its use in routine clinical practice requires the validation through controlled clinical trials. In addition the collection, administration and control of plasma is technically demanding and needs a clear support before broadly recommending it. Different scientific institutions and international organisms had clearly suggested to prioritize the application of novel therapeutic techniques with yet unproven efficacy within the context of clinical studies over its empirical use.

On the other hand, for the present study, intervention strategy is proposed in "add-on" modality over the antiviral treatment that each participant may be already receiving, since they represent completely different therapeutic approaches. As such, participation in the present study will not condition the possibility of the participants to receive other treatments, either in intervention or control arms.

4. Study objectives Primary objective Analyze the difference between arms on an ordinal score of six mutually exclusive categories at day 30 after study initiation. This score includes the following categories

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Covid-19 through qualitative polymerase-reverse transcriptase (qRT-PCR -GeneDX Co, Ltd o similar).
* Imagining-diagnosed pneumonia (Rx or CT scan).
* MSOFA score (Modified SOFA) of 2 or more (modified organic failure assessment)
* Informed consent.

Exclusion Criteria:

* Pregnant women
* Women at reproductive age not willing to avoid unprotected sexual intercourse up to Day 30 after study initiation.
* Women in the breastfeeding period
* Patients receiving experimental treatments under development within 30 days prior to study initiation.
* Patients with a previous history of allergic reactions to blood or blood-components transfusion.
* Diagnosis or clinical suspicion of an alternative microbiological cause for pneumonia besides COVID-19
* Use of systemic corticosteroids within 15 days prior to entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-09-27 (Actual); Study Completion 2020-09-27 (Actual)

PRIMARY OUTCOMES:
Clinical status during follow-up at 30th day | 30th Day since study preparation infusion (Placebo or Convalescent SARS COVID-19 plasma)
  Ordinal outcome with six mutually exclusive categories to describe the patient's clinical status during follow-up. The six categories are: (1) death; (2) in intensive care; (3) hospitalised but requiring supplemental oxygen; (4) hospitalised and not requiring supplemental oxygen; (5) discharged but unable to resume normal activities; or (6) discharged with full resumption of normal activities.

SECONDARY OUTCOMES:
Clinical status during follow-up at 7th day | 7th Day since study preparation infusion (Placebo or Convalescent SARS COVID-19 plasma)
  Ordinal outcome with six mutually exclusive categories to describe the patient's clinical status during follow-up. The six categories are: (1) death; (2) in intensive care; (3) hospitalised but requiring supplemental oxygen; (4) hospitalised and not requiring supplemental oxygen; (5) discharged but unable to resume normal activities; or (6) discharged with full resumption of normal activities.
Clinical status during follow-up at 14th day | 14th Day since study preparation infusion (Placebo or Convalescent SARS COVID-19 plasma)
  Ordinal outcome with six mutually exclusive categories to describe the patient's clinical status during follow-up. The six categories are: (1) death; (2) in intensive care; (3) hospitalised but requiring supplemental oxygen; (4) hospitalised and not requiring supplemental oxygen; (5) discharged but unable to resume normal activities; or (6) discharged with full resumption of normal activities.
Time until hospital discharge (days). | Whenever the patient is discharge from the hospital or die without discharge, through study completion, an average of 14 days from admission
  Hospital discharge or intrahospital death
Time until discharge from ICU (days) | Whenever the patient is discharge from ICU or die in ICU, through study completion, an average of 10 days from admission
  ICU discharge or ICU death
Time to death | In a 30 days follow up period
  Death and time to death
Time until complete functional recovery | Whenever the patient returns to basal functional status until 1 month from discharge
  Time until complete functional recovery (according to basal status).
Percentage of participants with adverse events / serious adverse events | In a 30 days follow up period
  Percentage of participants with adverse events / serious adverse events
Percentage of patients with negative SARS-CoV-3 PCR at Day 14th | 14th Day since study preparation infusion (Placebo or Convalescent SARS COVID-19 plasma)
  Percentage of patients with negative SARS-CoV-3 PCR
D Dimer plasma concentration at Day 14th | 14th Day since study preparation infusion (Placebo or Convalescent SARS COVID-19 plasma)
  D Dimer plasma concentration
Ferritin plasma concentration at Day 13th | 13th Day since study preparation infusion (Placebo or Convalescent SARS COVID-19 plasma)
  Ferritin plasma concentration
Plasma concentration of neutralizing antibodies at Day 2nd | 2nd Day since study preparation infusion (Placebo or Convalescent SARS COVID-19 plasma)
  Plasma concentration of neutralizing antibodies
Plasma concentration of neutralizing antibodies at Day 7th | 7th Day since study preparation infusion (Placebo or Convalescent SARS COVID-19 plasma)
  Plasma concentration of neutralizing antibodies
Post-transfusion adverse reactions | In a 30 days follow up period
  Post-transfusion adverse reactions between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Nora A Fuentes, MD, Principal Investigator — Hospital Privado de la Comunidad de Mar del Plata; Florencia Otermin, MD, Principal Investigator — Hospital Italiano de la Plata; Esteban Nannini, MD, Principal Investigator — Sanatorio Britanico Rosario, pcia Santa Fe; Karina Rainiero, MD, Principal Investigator — Suiza Argentina; Erica Miyazaki, MD, Principal Investigator — Clinica Zabala; Gabriela Vidiella, MD, Principal Investigator — Sanatorio Agote; Wanda Cornistein, MD, Principal Investigator — Austral University, Argentina; Leandro Burgos, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maiztegui JI, Fernandez NJ, de Damilano AJ. Efficacy of immune plasma in treatment of Argentine haemorrhagic fever and association between treatment and a late neurological syndrome. Lancet. 1979 Dec 8;2(8154):1216-7. doi: 10.1016/s0140-6736(79)92335-3. PMID 92624
- [Background] Tanne JH. Covid-19: FDA approves use of convalescent plasma to treat critically ill patients. BMJ. 2020 Mar 26;368:m1256. doi: 10.1136/bmj.m1256. No abstract available. PMID 32217555
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Roback JD, Guarner J. Convalescent Plasma to Treat COVID-19: Possibilities and Challenges. JAMA. 2020 Apr 28;323(16):1561-1562. doi: 10.1001/jama.2020.4940. No abstract available. PMID 32219429
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Kalil AC. Treating COVID-19-Off-Label Drug Use, Compassionate Use, and Randomized Clinical Trials During Pandemics. JAMA. 2020 May 19;323(19):1897-1898. doi: 10.1001/jama.2020.4742. No abstract available. PMID 32208486
- [Background] Angus DC. Optimizing the Trade-off Between Learning and Doing in a Pandemic. JAMA. 2020 May 19;323(19):1895-1896. doi: 10.1001/jama.2020.4984. No abstract available. PMID 32227198
- [Result] Luke TC, Kilbane EM, Jackson JL, Hoffman SL. Meta-analysis: convalescent blood products for Spanish influenza pneumonia: a future H5N1 treatment? Ann Intern Med. 2006 Oct 17;145(8):599-609. doi: 10.7326/0003-4819-145-8-200610170-00139. Epub 2006 Aug 29. PMID 16940336
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Simonovich VA, Burgos Pratx LD, Scibona P, Beruto MV, Vallone MG, Vazquez C, Savoy N, Giunta DH, Perez LG, Sanchez MDL, Gamarnik AV, Ojeda DS, Santoro DM, Camino PJ, Antelo S, Rainero K, Vidiella GP, Miyazaki EA, Cornistein W, Trabadelo OA, Ross FM, Spotti M, Funtowicz G, Scordo WE, Losso MH, Ferniot I, Pardo PE, Rodriguez E, Rucci P, Pasquali J, Fuentes NA, Esperatti M, Speroni GA, Nannini EC, Matteaccio A, Michelangelo HG, Follmann D, Lane HC, Belloso WH; PlasmAr Study Group. A Randomized Trial of Convalescent Plasma in Covid-19 Severe Pneumonia. N Engl J Med. 2021 Feb 18;384(7):619-629. doi: 10.1056/NEJMoa2031304. Epub 2020 Nov 24. PMID 33232588